CLINICAL TRIAL: NCT02365922
Title: Rare Diseases Clinical Research Network Advancing Research and Treatment for Frontotemporal Lobar Degeneration [ARTFL]: Research Projects 1 & 2
Brief Title: Advancing Research and Treatment for Frontotemporal Lobar Degeneration (ARTFL)
Acronym: ARTFL
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The Bluefield Project to Cure Frontotemporal Dementia (Other); Tau Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: ARTFL8101; 1U54NS092089-01 (NIH)
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: FTLD; Progressive Supranuclear Palsy (PSP); Frontotemporal Dementia (FTD); Corticobasal Degeneration (CBD); PPA Syndrome; Behavioral Variant Frontotemporal Dementia (bvFTD); Semantic Variant Primary Progressive Aphasia (svPPA); Nonfluent Variant Primary Progressive Aphasia (nfvPPA); FTD With Amyotrophic Lateral Sclerosis (FTD/ALS); Amyotrophic Lateral Sclerosis (ALS); Oligosymptomatic PSP (oPSP); Corticobasal Syndrome (CBS)
Keywords: FTLD, PSP, CBD, PPA, FTD, FTD-ALS, CBS, ALS, svPPA, nfvPPA, oPSP
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Supranuclear Palsy, Progressive; Frontotemporal Dementia; Corticobasal Degeneration; Primary Progressive Nonfluent Aphasia; Amyotrophic Lateral Sclerosis; Color Vision Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, cell lines and cerebrospinal fluid will be retained by study investigators and stored at NIH-funded repositories.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with FTLD or family members: Participants with FTLD syndrome diagnoses and/or strong family histories of FTLD.

SUMMARY:
Frontotemporal Lobar Degeneration (FTLD) is the neuropathological term for a collection of rare neurodegenerative diseases that correspond to four main overlapping clinical syndromes: frontotemporal dementia (FTD), primary progressive aphasia (PPA), corticobasal degeneration syndrome (CBS) and progressive supranuclear palsy syndrome (PSPS). The goal of this study is to build a FTLD clinical research consortium to support the development of FTLD therapies for new clinical trials. The consortium, referred to as Advancing Research and Treatment for Frontotemporal Lobar Degeneration (ARTFL), will be headquartered at UCSF and will partner with six patient advocacy groups to manage the consortium. Participants will be evaluated at 14 clinical sites throughout North America and a genetics core will genotype all individuals for FTLD associated genes.

DETAILED DESCRIPTION:
Frontotemporal Lobar Degeneration (FTLD) is the neuropathological term for a collection of rare neurodegenerative diseases that correspond to four main overlapping clinical syndromes: frontotemporal dementia (FTD), primary progressive aphasia (PPA), corticobasal degeneration syndrome (CBS) and progressive supranuclear palsy syndrome (PSPS). The goal of this study is to build a FTLD clinical research consortium (FTLD CRC) to support the development of FTLD therapies for new clinical trials. The FTLD CRC will be headquartered at UCSF and will partner with six patient advocacy groups to manage the consortium. Patients will be evaluated at 13 clinical sites throughout North America and a genetics core will genotype all individuals for FTLD associated genes.

The study will be divided into 2 projects. The first project will be Preparing for Sporadic FTLD Clinical Trials and the second project will be a Longitudinal Assessment of Familial FTLD. Self-registration for an online registry will be available for patients and families with any FTLD syndrome. Eligible participants for research Projects 1 and 2 FTLD will be invited to a CRC site for clinical evaluations. All enrolled participants in both research projects will have a site visit consisting of a neurological exam, medical and family history, cognitive testing, and a blood draw.

Participants in Project 1 who have a diagnosis of Progressive Supranuclear Palsy Syndrome will have two additional assessments. A lumbar puncture (LP) will be performed for CSF collection, and an MRI scan of the brain will be done.

Participants in Project 2: Longitudinal Assessment of familial FTLD will return for a follow-up visit in 12 months; procedures at the follow-up visit will be identical to those at baseline. Additionally, asymptomatic participants will undergo MRI scans at both visits.

ELIGIBILITY:
1. Inclusion Criteria:Must meet one of the following research diagnostic criteria for a Frontotemporal lobar degeneration (FTLD) syndrome: behavioral variant frontotemporal dementia (bvFTD), primary progressive aphasia (PPA), semantic variant primary progressive aphasia (svPPA), nonfluent variant primary progressive aphasia (nfvPPA), frontotemporal dementia with amyotrophic lateral sclerosis (FTD/ALS), amyotrophic lateral sclerosis alone, corticobasal syndrome (CBS), progressive supranuclear palsy (PSP) or oligosymptomatic PSP (oPSP), or have a strong family history of FTLD syndromes.
2. Between 18 and 85 (inclusive) years of age.
3. Able to walk (with assistance) at the time of enrollment.
4. Have a reliable study partner who can provide an independent evaluation of functioning.
5. Speak English or Spanish
6. Have Mini Mental State Exam (MMSE) scores between 15 - 30 (inclusive).

Exclusion Criteria:

1. Known presence of a structural brain lesion (e.g. tumor,cortical infarct) that could reasonably explain symptoms in a symptomatic participant without a known f-FTLD causing mutation.
2. Known presence of an Alzheimer's disease causing mutation in PSEN1, PSEN2 or APP; or neuropathological evidence for Alzheimer's disease as a cause of syndrome (from brain biopsy).
3. A previous history of Korsakoff encephalopathy, severe alcohol dependence (within 5 years of onset of dementia), frequent alcohol or other substance intoxication, or other neurological disorder (such as multiple sclerosis)
4. Evidence through history or laboratory testing of B12 deficiency (B12 < 95% of local laboratory's normal value), hypothyroidism (TSH >150% of normal), HIV positive,renal failure (creatinine > 2), liver failure (ALT or AST > two times normal), respiratory failure (requiring oxygen), extra-axial brain tumor (with visible compression of the brain parenchyma), large cerebral infarct that could account for clinical syndrome, large confluent white matter lesions (grades 3 or 4, [107] significant systemic medical illnesses such as deteriorating cardiovascular disease;
5. Current medication likely to affect CNS functions in the opinion of the site PI: long acting benzodiazepines such as diazepam (short-acting benzodiazepines are OK), non-SSRI antidepressants (SSRIs or trazodone are OK), no lithium, typical neuroleptics as listed in the Manual of Procedures, narcotics (codeine is OK, but hold 24 hours before neuropsychological testing), anticonvulsants (outside of therapeutic ranges), antihistamines (if taking greater than three times per week; hold 24 hours before neuropsychological testing).
6. In the site investigator's opinion, the participant cannot complete sufficient key study procedures, or equivalent assessment of impairment level.
7. For groups where MRI scans are planned procedures, any contraindication for MRI scanning, such as pacemaker or other implanted metals.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of a frontotemporal lobar degeneration (FTLD) syndrome, including progressive supranuclear palsy (PSP), semantic variant primary progressive aphasia (svPPA), and frontotemporal dementia with amyotrophic lateral sclerosis (FTD-ALS). Family members of patients with FTLD syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 1489 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Scores of UDS FTLD Module Tests | Baseline, 12 mo.
  Neuropsychological test scores from the Uniform Data Set FTLD Module will be collected and compared across patient populations.

SECONDARY OUTCOMES:
Progressive Supranuclear Palsy Rating Scale (PSPRS) | Baseline
  Scores will be compared among patient populations
Neuroimaging | Baseline; 12 months
  In asymptomatic family members of FTLD patients, changes from baseline neuroimaging will be assessed 12 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Boxer, MD, PhD, Principal Investigator — Study PI
Locations (17):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University Massachusetts General Hospital, Charlestown, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Case Western Reserve University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington Harborview Medical Center, Seattle, Washington
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Toronto, Toronto, Ontario

REFERENCES:
- [Background] Boxer AL, Knopman DS, Kaufer DI, Grossman M, Onyike C, Graf-Radford N, Mendez M, Kerwin D, Lerner A, Wu CK, Koestler M, Shapira J, Sullivan K, Klepac K, Lipowski K, Ullah J, Fields S, Kramer JH, Merrilees J, Neuhaus J, Mesulam MM, Miller BL. Memantine in patients with frontotemporal lobar degeneration: a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2013 Feb;12(2):149-56. doi: 10.1016/S1474-4422(12)70320-4. Epub 2013 Jan 2. PMID 23290598
- [Background] Boxer AL, Garbutt S, Seeley WW, Jafari A, Heuer HW, Mirsky J, Hellmuth J, Trojanowski JQ, Huang E, DeArmond S, Neuhaus J, Miller BL. Saccade abnormalities in autopsy-confirmed frontotemporal lobar degeneration and Alzheimer disease. Arch Neurol. 2012 Apr;69(4):509-17. doi: 10.1001/archneurol.2011.1021. PMID 22491196
- [Background] Boxer AL, Lang AE, Grossman M, Knopman DS, Miller BL, Schneider LS, Doody RS, Lees A, Golbe LI, Williams DR, Corvol JC, Ludolph A, Burn D, Lorenzl S, Litvan I, Roberson ED, Hoglinger GU, Koestler M, Jack CR Jr, Van Deerlin V, Randolph C, Lobach IV, Heuer HW, Gozes I, Parker L, Whitaker S, Hirman J, Stewart AJ, Gold M, Morimoto BH; AL-108-231 Investigators. Davunetide in patients with progressive supranuclear palsy: a randomised, double-blind, placebo-controlled phase 2/3 trial. Lancet Neurol. 2014 Jul;13(7):676-85. doi: 10.1016/S1474-4422(14)70088-2. Epub 2014 May 27. PMID 24873720
- [Background] Rosen HJ, Alcantar O, Zakrzewski J, Shimamura AP, Neuhaus J, Miller BL. Metacognition in the behavioral variant of frontotemporal dementia and Alzheimer's disease. Neuropsychology. 2014 May;28(3):436-47. doi: 10.1037/neu0000012. Epub 2014 Feb 17. PMID 24548124
- [Background] Rosen HJ, Alcantar O, Rothlind J, Sturm V, Kramer JH, Weiner M, Miller BL. Neuroanatomical correlates of cognitive self-appraisal in neurodegenerative disease. Neuroimage. 2010 Feb 15;49(4):3358-64. doi: 10.1016/j.neuroimage.2009.11.041. Epub 2009 Dec 1. PMID 19961939
- [Background] Rohrer JD, Rosen HJ. Neuroimaging in frontotemporal dementia. Int Rev Psychiatry. 2013 Apr;25(2):221-9. doi: 10.3109/09540261.2013.778822. PMID 23611351
- [Background] Boeve BF. Progressive supranuclear palsy. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1:S192-4. doi: 10.1016/S1353-8020(11)70060-8. PMID 22166432
- [Background] Boeve BF. The multiple phenotypes of corticobasal syndrome and corticobasal degeneration: implications for further study. J Mol Neurosci. 2011 Nov;45(3):350-3. doi: 10.1007/s12031-011-9624-1. Epub 2011 Aug 19. PMID 21853287
- [Derived] Tipton PW, Deutschlaender AB, Savica R, Heckman MG, Brushaber DE, Dickerson BC, Gavrilova RH, Geschwind DH, Ghoshal N, Graff-Radford J, Graff-Radford NR, Grossman M, Hsiung GR, Huey ED, Irwin DJ, Jones DT, Knopman DS, McGinnis SM, Rademakers R, Ramos EM, Forsberg LK, Heuer HW, Onyike C, Tartaglia C, Domoto-Reilly K, Roberson ED, Mendez MF, Litvan I, Appleby BS, Grant I, Kaufer D, Boxer AL, Rosen HJ, Boeve BF, Wszolek ZK; ALLFTD Consortium. Differences in Motor Features of C9orf72, MAPT, or GRN Variant Carriers With Familial Frontotemporal Lobar Degeneration. Neurology. 2022 Sep 13;99(11):e1154-e1167. doi: 10.1212/WNL.0000000000200860. Epub 2022 Jul 5. PMID 35790423
- [Derived] Gendron TF, Heckman MG, White LJ, Veire AM, Pedraza O, Burch AR, Bozoki AC, Dickerson BC, Domoto-Reilly K, Foroud T, Forsberg LK, Galasko DR, Ghoshal N, Graff-Radford NR, Grossman M, Heuer HW, Huey ED, Hsiung GR, Irwin DJ, Kaufer DI, Leger GC, Litvan I, Masdeu JC, Mendez MF, Onyike CU, Pascual B, Ritter A, Roberson ED, Rojas JC, Tartaglia MC, Wszolek ZK, Rosen H, Boeve BF, Boxer AL; ALLFTD consortium; Petrucelli L. Comprehensive cross-sectional and longitudinal analyses of plasma neurofilament light across FTD spectrum disorders. Cell Rep Med. 2022 Apr 19;3(4):100607. doi: 10.1016/j.xcrm.2022.100607. eCollection 2022 Apr 19. PMID 35492244
- [Derived] Rojas JC, Wang P, Staffaroni AM, Heller C, Cobigo Y, Wolf A, Goh SM, Ljubenkov PA, Heuer HW, Fong JC, Taylor JB, Veras E, Song L, Jeromin A, Hanlon D, Yu L, Khinikar A, Sivasankaran R, Kieloch A, Valentin MA, Karydas AM, Mitic LL, Pearlman R, Kornak J, Kramer JH, Miller BL, Kantarci K, Knopman DS, Graff-Radford N, Petrucelli L, Rademakers R, Irwin DJ, Grossman M, Ramos EM, Coppola G, Mendez MF, Bordelon Y, Dickerson BC, Ghoshal N, Huey ED, Mackenzie IR, Appleby BS, Domoto-Reilly K, Hsiung GR, Toga AW, Weintraub S, Kaufer DI, Kerwin D, Litvan I, Onyike CU, Pantelyat A, Roberson ED, Tartaglia MC, Foroud T, Chen W, Czerkowicz J, Graham DL, van Swieten JC, Borroni B, Sanchez-Valle R, Moreno F, Laforce R, Graff C, Synofzik M, Galimberti D, Rowe JB, Masellis M, Finger E, Vandenberghe R, de Mendonca A, Tagliavini F, Santana I, Ducharme S, Butler CR, Gerhard A, Levin J, Danek A, Otto M, Sorbi S, Cash DM, Convery RS, Bocchetta M, Foiani M, Greaves CV, Peakman G, Russell L, Swift I, Todd E, Rohrer JD, Boeve BF, Rosen HJ, Boxer AL; ALLFTD and GENFI consortia. Plasma Neurofilament Light for Prediction of Disease Progression in Familial Frontotemporal Lobar Degeneration. Neurology. 2021 May 4;96(18):e2296-e2312. doi: 10.1212/WNL.0000000000011848. Epub 2021 Apr 7. PMID 33827960